CLINICAL TRIAL: NCT04170010
Title: Postprandial Gut Hormone Responses and Meal-induced Thermogenesis After Non-surgical Long-term Weight Loss; Comparison With Surgically Treated Obese Individuals
Brief Title: Long Term Effects of Weight Loss on Post-prandial Gut Hormone Responses and Meal Induced Thermogenesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Alexandros Kokkinos, Associate Professor in Internal Medicine, National and Kapodistrian University of Athens
Other Study IDs: Weight loss gut peptide study
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Morbid Obesity
Keywords: Weight loss; Gut peptides; Meal-induced thermogenesis; Glycemia
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conservatively managed group: Individuals with conservatively managed obesity
- Surgically managed group: Individuals with a past history of bariatric surgery (Roux-en-Y gastric bypass/Sleeve gastrectomy) for the management of obesity

SUMMARY:
A study to examine post-prandial gut-hormone secretion, meal-induced thermogenesis, fasting plasma metabolomic/lipidomic and cardiovascular indices among surgically managed obese individuals in the long term compared to conservatively managed obese patients.

DETAILED DESCRIPTION:
This is a protocol for the study of post-prandial gut peptide response and meal-induced thermogenesis in a group of 15 conservatively managed (through diet and exercise) morbidly obese individuals. During two separate visits in the study site, anthropometric and bioelectric impendence data will be collected, resting metabolic rate will be measured, and the patients will undergo a panel of cardiovascular examinations (heart rate variability, baroreflex sensitivity, heart ultrasound). On a separate occasion, they will consume a standardized test mixed meal and complete visual analog scales for the subjective assessment of hunger and fullness every 30 minutes for 3 hours. At the same time points, blood samples will be collected for the consequent measurement of glucose, insulin, lipids, and gastrointestinal hormones. Additionally, immediately before and at 60', 120', 180' after the start of the consumption of the test meal, the resting metabolic rate of each participant will be assessed through indirect calorimetry, to quantify meal-induced thermogenesis. The observed induction of satiety and suppression of hunger, post prandial gut-peptide mobilization and change in metabolic rate will be compared to those of participants of trial no NCT03851874 (Morbidly obese patients that have undergone either Roux en Y gastric bypass or sleeve gastrectomy and participated in trial NCT03851874). Participants in the aforementioned cohort have been already followed-up during the first postoperative year and will attend the study site for another follow-up visit approximately 10 years postoperatively, whereby the same diagnostic evaluation described above will take place. Data analysis will take place within the bariatric cohort (longitudinal analysis of the effects of surgery and surgery types on anthropometric parameters, fasting and postprandial glycemia and lipemia, fasting NMR-Metabolomic/Lipidomic profiles, Indices of insulin resistance, echocardiography, energy expenditure) as well as between the two groups in a cross-sectional manner.

ELIGIBILITY:
Inclusion Criteria:

* For the conservatively managed cohort:

  1. Morbid obesity based on BMI > 40kg/m2, managed exclusively with conservative measures (hypocaloric diet and/or increased physical activity and/or behavioral therapy)
  2. Age between 18 and 65 years
* For the bariatric cohort: Participation in NCT03851874 trial

Exclusion Criteria:

1. Serious and life threatening comorbidities (renal, cardiac, liver failure, or malignancy)
2. Alcohol or other substance abuse
3. Use of licenced or off-label weight loss medications during the past 6 months
4. Concurrent psychiatric illness
5. Known history of diabetes mellitus (remitted cases excluded)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intervention group: participants of NCT03851874 trial Control group: conservatively (non-surgically, non-pharmaceutically) managed obese individuals among ambulatory patients of the obesity outpatient clinic of the 1st Department of Propaedeutic Internal Medicine ("Laiko" General Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in postprandial Gut peptide (ghrelin, Gastric Inhibitory Peptide, Secretin, Peptide Tyrosine-Tyrosine - , Glucagon-like peptide - 1, Oxyntomodulin, Glicentin) responses | 8-10 years following primary weight-loss intervention
  Change in the cumulative postprandial response for the aforementioned gut hormones
Change in weight, fat mass and lean body mass | 8-10 years following primary weight-loss intervention
  Change in weight (percentage of weight following each intervention)

SECONDARY OUTCOMES:
Change in postprandial glycemia | 8-10 years following primary weight-loss intervention
  Change in postprandial glycemia
Change in postprandial insulinemia | 8-10 years following primary weight-loss intervention
  Change in the cumulative postprandial response for insulin
Change in postprandial triglyceridemia | 8-10 years following primary weight-loss intervention
  Change in the cumulative postprandial response for triglycerides
Change in Insulin resistance | 8-10 years following primary weight-loss intervention
  Change in Insulin resistance indices (HOMA-R, MMTT-derived Matsuda index)
Change in serum metabolomic and lipidomic parameters | 8-10 years following primary weight-loss intervention
  Change in levels of lipoprotein clusters, branched-chain amino-acids, LDL/HDL-Subtypes, Trimethylamine N-oxide assessed by NMR spectroscopy
Change in resting metabolic rate following meal ingestion | 8-10 years following primary weight-loss intervention
  Change in the cumulative postprandial thermogenesis
Change in fasting serum adipokines | 8-10 years following primary weight-loss intervention
  Change of fasting leptin, adiponektin concentrations
Change in fasting plasma Activins and follistatins | 8-10 years following primary weight-loss intervention
  Change in fasting plasma Activin A, B, AB, follistatin and follistatin-like 3
Change in postprandial Visual Analog Scale scores for hunger and satiety | 8-10 years following primary weight-loss intervention
  Change in postprandial areas under the curve of subjective hunger and satiety expressed in Visual Analog Scales

OTHER OUTCOMES:
Change in baroreflex sensitivity | 8-10 years following primary weight-loss intervention
  Changes in baroreflex sensitivity
Change in heart rate variability | 8-10 years following primary weight-loss intervention
  Changes in heart rate variability
Change in aortic distensibility | 8-10 years following primary weight-loss intervention
  Aortic distensibility will be evaluated by calculating the systolic and diastolic aortic diameter through M-mode echocardiography, 3 cm above the aortic valve, using the formula described in reference no 4 (PMID: 2282929)
Change in echocardiographic cardiac phenotype | 8-10 years following primary weight-loss intervention
  Change in echocardiographic cardiac structural indices and measures of systolic and diastolic function

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Kokkinos, MD, PhD, Principal Investigator — First Department of Propaedeutic Medicine, NKUA
Locations (1):
- Diabetes Clinical Research Laboratory, 1st Department of Propaedeutic Internal Medicine, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perakakis N, Kokkinos A, Peradze N, Tentolouris N, Ghaly W, Pilitsi E, Upadhyay J, Alexandrou A, Mantzoros CS. Circulating levels of gastrointestinal hormones in response to the most common types of bariatric surgery and predictive value for weight loss over one year: Evidence from two independent trials. Metabolism. 2019 Dec;101:153997. doi: 10.1016/j.metabol.2019.153997. Epub 2019 Oct 28. PMID 31672446
- [Background] Liaskos C, Koliaki C, Alexiadou K, Argyrakopoulou G, Tentolouris N, Diamantis T, Alexandrou A, Katsilambros N, Kokkinos A. Roux-en-Y Gastric Bypass Is More Effective than Sleeve Gastrectomy in Improving Postprandial Glycaemia and Lipaemia in Non-diabetic Morbidly Obese Patients: a Short-term Follow-up Analysis. Obes Surg. 2018 Dec;28(12):3997-4005. doi: 10.1007/s11695-018-3454-y. PMID 30112599
- [Background] Yousseif A, Emmanuel J, Karra E, Millet Q, Elkalaawy M, Jenkinson AD, Hashemi M, Adamo M, Finer N, Fiennes AG, Withers DJ, Batterham RL. Differential effects of laparoscopic sleeve gastrectomy and laparoscopic gastric bypass on appetite, circulating acyl-ghrelin, peptide YY3-36 and active GLP-1 levels in non-diabetic humans. Obes Surg. 2014 Feb;24(2):241-52. doi: 10.1007/s11695-013-1066-0. PMID 23996294
- [Background] Stefanadis C, Stratos C, Boudoulas H, Kourouklis C, Toutouzas P. Distensibility of the ascending aorta: comparison of invasive and non-invasive techniques in healthy men and in men with coronary artery disease. Eur Heart J. 1990 Nov;11(11):990-6. doi: 10.1093/oxfordjournals.eurheartj.a059639. PMID 2282929
- [Derived] Kokkinos A, Tsilingiris D, Simati S, Stefanakis K, Angelidi AM, Tentolouris N, Anastasiou IA, Connelly MA, Alexandrou A, Mantzoros CS. Bariatric surgery, through beneficial effects on underlying mechanisms, improves cardiorenal and liver metabolic risk over an average of ten years of observation: A longitudinal and a case-control study. Metabolism. 2024 Mar;152:155773. doi: 10.1016/j.metabol.2023.155773. Epub 2024 Jan 3. PMID 38181882
- [Derived] Stefanakis K, Kokkinos A, Simati S, Argyrakopoulou G, Konstantinidou SK, Kouvari M, Kumar A, Kalra B, Mantzoros CS. Circulating levels of all proglucagon-derived peptides are differentially regulated postprandially by obesity status and in response to high-fat meals vs. high-carbohydrate meals. Clin Nutr. 2023 Aug;42(8):1369-1378. doi: 10.1016/j.clnu.2023.06.026. Epub 2023 Jun 28. PMID 37418844